CLINICAL TRIAL: NCT06542406
Title: Can the Fluctuation Observed in the Endotracheal Tube With Compression Applied to the Epigastric Region be Used as a Confirmation Method for Endotracheal Intubation?
Brief Title: Can Endotracheal Tube Fluctuation With Epigastric Compression Be Used as a Confirmation Method for Endotracheal Intubation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, kudret selki, Researcher Assistant in Emergency Department, Duzce University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DuzceUniversityEM
Record Dates: First submitted 2024-07-26; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Intubation, Intratracheal
Keywords: endotracheal intubation; esophageal placement; epigastric fluctuation
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Endotracheal intubation (Other): Patients admitted to the emergency department between 01/05/2021 and 30/05/2022, who were older than 18 years of age and who underwent ETE outside the hospital or within the first hour of arrival to the emergency department were included in the study.
  Interventions: Device: Endotracheal intubation

INTERVENTIONS:
Device: Endotracheal intubation — The first 40 successful and the first 40 unsuccessful ETE procedures were included in the study.

SUMMARY:
Endotracheal intubation (ETE) may also need to be performed outside the hospital as advanced airway management. In such cases, facilities such as imaging methods, ultrasound or capnography may not be available and only traditional methods such as auscultation of lung sounds, auscultation of the epigastric region without hearing airflow, observation of chest expansion after ventilation, observation of water vapor in the tube may have to be used. Despite all these observational methods and equipment used, it is recommended to keep in mind that there may be errors and to try to provide confirmation with more than one method.

Especially in disaster situations where technological infrastructure is not available and sometimes outside the hospital, the use of traditional methods based on examination may be of vital importance. The traditional methods mentioned above are mostly used to detect tracheal localization and to exclude esophageal localization. In our observations in patients with cardiopulmonary arrest, the investigators noticed that in the case of esophageal placement of the tube, manual compression of the epigastric region produced a fluctuation in the tube and valved balloon caused by airflow. The investigators thought that this could be a method to confirm esophageal placement. The aim of this study was to investigate the usefulness of epigastric manual compression in the confirmation of esophageal placement of the tube.

DETAILED DESCRIPTION:
Patients who underwent ETE outside the hospital or in the first hour of arrival to the emergency department were evaluated after the procedure. Out-of-hospital ETE was performed by experienced paramedics working in the emergency ambulance service, and ETE in the emergency department was performed by emergency medicine residents or emergency medicine specialists with at least 2 years of emergency department experience. Out-of-hospital procedures were performed at the first visit to the emergency department, and procedures performed in the emergency department were confirmed by ETE immediately after the procedure.

Confirmation was performed single-blind by emergency medicine specialists with at least 5 years of experience, without knowing who performed the procedure and where (in or out of the hospital). Confirmation was performed by auscultation of lung sounds (from the anterior and lateral sides of both lungs, upper and lower zones), evaluation of equal participation of both thoraxes in breathing by inspection, auscultation of the epigastric region, placement of capnography, monitoring of water vapor in the tube, manual compression of the epigastric region at least three times and evaluation of fluctuation in the tube, and pulse oximetry monitoring.

Epigastric compression was performed by applying pressure to the epigastric region at least three times with the volar side of the intubated patient while the patient was ventilated with a balloon-valved mask. During this procedure, the fluctuation of the air and fluid in the stomach inside the esophageal tube can be observed and its sound can be heard. It can be applied from the first inhalation.

The ultrasonography (USG) procedure was evaluated by placing a linear ultrasound probe [SonoSite M-Turbo linear probe (13-6 MHz), Sonosite, Inc, Bothell, WA, USA] in the transverse position on the anterior side of the neck, just above the suprasternal notch, and observing the position of the tube (presence of a double path sign) and pleural sliding movement. While a single semicircular echogenic area is observed when the tube is in the trachea, a second semicircular echogenic area is observed when the tube is located in the esophagus. USG was performed immediately after the ETE procedure. In patients in whom double pathway sign was observed and pleural sliding motion was not observed, the patient was re-intubated by the experienced specialist performing USG. It was confirmed by USG again. These procedures were categorized as "failed".

partial endtidal carbon dioxide (PETCO2) measurement by capnography was performed using a mainstream EMMA® Capnograph (PHASEIN AB Svärdvägen, Danderyd, Sweden) for intubated patients. It was assessed by the detection of PETCO2 greater than 5 mmHg after five breaths and the appearance of a typical square waveform.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age
* Underwent ETE outside the hospital or within the first hour of arrival to the emergency department

Exclusion Criteria:

* Patients in whom ETE was previously confirmed by USG or PETCO2,
* Patients intubated at external centers
* Patients who had known airway stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-03-04 (Actual)

PRIMARY OUTCOMES:
Confirmation with ultrasonography: Successful or Failed | 13 months
  Fluctuation with Epigastric Compression: Yes or No
  Failed Successful Failed

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Boğan, MD, Study Director — Duzce University, School of Medicine, Emergency Department
Locations (1):
- Duzce University, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data can be shared with those who request it.

REFERENCES:
- [Result] Farrokhi M, Yarmohammadi B, Mangouri A, Hekmatnia Y, Bahramvand Y, Kiani M, Nasrollahi E, Nazari-Sabet M, Manoochehri-Arash N, Khurshid M, Mosalanejad S, Hajizadeh V, Amani-Beni R, Moallem M, Farahmandsadr M. Screening Performance Characteristics of Ultrasonography in Confirmation of Endotracheal Intubation; a Systematic Review and Meta-analysis. Arch Acad Emerg Med. 2021 Oct 26;9(1):e68. doi: 10.22037/aaem.v9i1.1360. eCollection 2021. PMID 34870234
- [Result] Li X, Zhang J, Karunakaran M, Hariharan VS. Diagnostic accuracy of ultrasonography for the confirmation of endotracheal tube intubation: a systematic review and meta-analysis. Med Ultrason. 2023 Mar 30;25(1):72-81. doi: 10.11152/mu-3594. Epub 2022 Jun 3. PMID 36780595
- [Result] Kramer-Johansen J, Dorph E, Steen PA. Detection of carbon dioxide in expired air after oesophageal intubation; the role of bystander mouth-to-mouth ventilation. Acta Anaesthesiol Scand. 2008 Jan;52(1):155-7. doi: 10.1111/j.1399-6576.2007.01503.x. Epub 2007 Nov 12. PMID 17999713

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/06/NCT06542406/Prot_SAP_000.pdf